CLINICAL TRIAL: NCT00365170
Title: A Randomised, Parallel-group, Open-label, Multinational Trial Comparing the Safety and Efficacy of Insulin Aspart (NovoRapid®) Versus Human Insulin (Actrapid®), Used in a Multiple Injection Regimen, in the Treatment of Pregnant Women With Type 1 Diabetes, Focusing on Maternal Hypoglycaemia and Pregnancy Outcomes
Brief Title: Efficacy and Safety of Insulin Aspart vs. Human Insulin During Pregnancy by Women With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1474
Record Dates: First submitted 2006-08-10; First posted 2006-08-17 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: human insulin
Drug: insulin aspart

SUMMARY:
This trial was conducted in Europe, Middle East, North America and South America.

The aim of this trial was to compare the use of an intensified insulin treatment with insulin aspart (NovoRapid®) versus human insulin (Actrapid®) in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Treated with insulin for at least 12 months
* Either plan to become pregnant in the immediate future, willing to undertake pre pregnancy counselling, and has a screening HbA1c lesser than or equal to 12.0%, or
* Pregnant with normal singleton pregnancy, gestational age for at least 10 weeks at the time of randomisation, confirmed by ultrasound scan.

Exclusion Criteria:

* Previous birth of child with a major congenital malformation
* More than 2 previous multiple miscarriages or stillbirths
* Severe hyperemesis gravidarum, requiring hospitalisation, according to Investigator judgement
* Subjects being treated for infertility
* Proliferative retinopathy or maculopathy requiring acute treatment
* Drug or alcohol abuse
* Impaired renal, hepatic or cardiac function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2002-09; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Relative risk of major maternal hypoglycaemia | after 24 hours

SECONDARY OUTCOMES:
Relative risk of major and minor hypoglycaemia
Diabetic complications
Obstetric complications
Other Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (1452, GCR), Study Director — Novo Nordisk A/S
Locations (87):
- Argentina (2):
  - Novo Nordisk Investigational Site, Ciudad de Buenos Aires
  - Novo Nordisk Investigational Site, Pcia de Cordoba
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Canada (6):
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Ottawa
  - Novo Nordisk Investigational Site, St. John's
  - Novo Nordisk Investigational Site, Toronto
  - Novo Nordisk Investigational Site, Vancouver
  - Novo Nordisk Investigational Site, Winnipeg
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Denmark (2):
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, København Ø
- Finland (3):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
- France (13):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Avignon
  - Novo Nordisk Investigational Site, Bondy
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Marseille Cédex 05
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Puyricard
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Valenciennes
- Novo Nordisk Investigational Site, Berlin, Germany
- Novo Nordisk Investigational Site, Athens, Greece
- Novo Nordisk Investigational Site, Dublin, Ireland
- Israel (4):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Petah Tikva
- Netherlands (7):
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Brunssum
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Roermond
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Utrecht
- Norway (3):
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Tromsø
  - Novo Nordisk Investigational Site, Trondheim
- Poland (8):
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Olsztyn
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Spain (4):
  - Novo Nordisk Investigational Site, Alicante
  - Novo Nordisk Investigational Site, Girona
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Seville
- United Kingdom (25):
  - Novo Nordisk Investigational Site, Ashington
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Edgbaston, Birmingham
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Norfolk
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Reading
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Southampton
  - Novo Nordisk Investigational Site, Stourbridge
  - Novo Nordisk Investigational Site, Worcester

REFERENCES:
- [Result] Mathiesen ER, Kinsley B, Amiel SA, Heller S, McCance D, Duran S, Bellaire S, Raben A; Insulin Aspart Pregnancy Study Group. Maternal glycemic control and hypoglycemia in type 1 diabetic pregnancy: a randomized trial of insulin aspart versus human insulin in 322 pregnant women. Diabetes Care. 2007 Apr;30(4):771-6. doi: 10.2337/dc06-1887. PMID 17392539
- [Result] Hod M, Jovanovic L. Improving outcomes in pregnant women with type 1 diabetes. Diabetes Care. 2007 Jul;30(7):e62. doi: 10.2337/dc07-0488. No abstract available. PMID 17596485
- [Result] Hod M, Damm P, Kaaja R, Visser GH, Dunne F, Demidova I, Hansen AS, Mersebach H; Insulin Aspart Pregnancy Study Group. Fetal and perinatal outcomes in type 1 diabetes pregnancy: a randomized study comparing insulin aspart with human insulin in 322 subjects. Am J Obstet Gynecol. 2008 Feb;198(2):186.e1-7. doi: 10.1016/j.ajog.2007.08.005. Epub 2007 Oct 1. PMID 17905178
- [Result] McCance DR, Damm P, Mathiesen ER, Hod M, Kaaja R, Dunne F, Jensen LE, Mersebach H. Evaluation of insulin antibodies and placental transfer of insulin aspart in pregnant women with type 1 diabetes mellitus. Diabetologia. 2008 Nov;51(11):2141-3. doi: 10.1007/s00125-008-1120-y. Epub 2008 Aug 23. No abstract available. PMID 18726086
- [Result] Heller S, Damm P, Mersebach H, Skjoth TV, Kaaja R, Hod M, Duran-Garcia S, McCance D, Mathiesen ER. Hypoglycemia in type 1 diabetic pregnancy: role of preconception insulin aspart treatment in a randomized study. Diabetes Care. 2010 Mar;33(3):473-7. doi: 10.2337/dc09-1605. Epub 2009 Dec 10. PMID 20007944
- [Result] Damm P, Mersebach H, Rastam J, Kaaja R, Hod M, McCance DR, Mathiesen ER. Poor pregnancy outcome in women with type 1 diabetes is predicted by elevated HbA1c and spikes of high glucose values in the third trimester. J Matern Fetal Neonatal Med. 2014 Jan;27(2):149-54. doi: 10.3109/14767058.2013.806896. Epub 2013 Jun 20. PMID 23687948
- [Derived] Altschuler JA, Casella SJ, MacKenzie TA, Curtis KM. The effect of cinnamon on A1C among adolescents with type 1 diabetes. Diabetes Care. 2007 Apr;30(4):813-6. doi: 10.2337/dc06-1871. PMID 17392542
- [Derived] Williams MM, Clouse RE, Nix BD, Rubin EH, Sayuk GS, McGill JB, Gelenberg AJ, Ciechanowski PS, Hirsch IB, Lustman PJ. Efficacy of sertraline in prevention of depression recurrence in older versus younger adults with diabetes. Diabetes Care. 2007 Apr;30(4):801-6. doi: 10.2337/dc06-1825. PMID 17392541
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com